CLINICAL TRIAL: NCT07282730
Title: Evaluation of Surgical Physicians' Awareness of Preoperative Patient Preparation
Brief Title: Awareness of Surgeons
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. Prof., Istinye University
Other Study IDs: 244-2025
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Awareness of Surgeon; Preoperative Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Surgeons' knowledge levels regarding preoperative evaluation — It aims to objectively reveal the current knowledge levels of surgical physicians, to increase their awareness, and to contribute to in-house training processes with the results obtained and to fill an important gap in the literature.

SUMMARY:
It aims to objectively reveal the current knowledge levels of surgical physicians, to increase their awareness, and to contribute to in-house training processes with the results obtained and to fill an important gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who voluntarily approved the participation form,
* Those who fully participated in the training and testing.

Exclusion Criteria:

* Those who did not complete the voluntary consent form,
* Those who did not participate in any phase of the training or testing,
* Participants with incomplete or inaccurate data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this study consists of all surgical specialists (both residents and specialists) working at Sultangazi Haseki Training and Research Hospital. The study will include physicians working in general surgery, orthopedics, neurosurgery, urology, ENT, and other surgical disciplines.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2025-12-17 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between pre- and post-training test scores (knowledge/awareness increase) | 1 hour
  The outcome is defined as the difference between the post-training and pre-training test scores assessing surgical awareness. Test scores range from 0 to 100, with higher scores indicating greater surgical awareness and knowledge. A positive difference reflects an increase in awareness following the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Gerber B, Roth EP, Laubach TA, De Jong L, Kasper TJ, Perry J, Johnson A, Krogman WL, Newton FA, Powell S, Bragg DA, Regehr J. Educating Family Physician Residents for Anesthetic Preoperative Evaluation and Assessment. Kans J Med. 2023 Sep 25;16(3):234-236. doi: 10.17161/kjm.vol16.20986. eCollection 2023. PMID 37791030
- [Result] Namara CM, O'Brien B, O'Reilly P. The learning experiences of student nurses in the perioperative environment: An integrative literature review. Nurse Educ Today. 2023 Dec;131:105985. doi: 10.1016/j.nedt.2023.105985. Epub 2023 Oct 9. PMID 37837917